CLINICAL TRIAL: NCT00073242
Title: Effects of Low-Dose Leptin on the Metabolic/Behavioral Phenotypes of the Formerly-Obese
Brief Title: Low-Dose Leptin and the Formerly-Obese
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 9631(completed)
Record Dates: First submitted 2003-11-18; First posted 2003-11-19 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Obesity
Keywords: leptin; obesity
MeSH Terms: conditions — Obesity | interventions — Leptin; Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- leptin repletion (Experimental): Repletion of leptin following weight loss induced by dietary modification.
  Interventions: Drug: Leptin; Behavioral: Dietary modification
- T3 repletion (Experimental): Repletion of T3 following weight loss induced by dietary modification.
  Interventions: Behavioral: Dietary modification; Drug: T3 repletion

INTERVENTIONS:
Drug: Leptin — leptin administration
  Other Names: no other names
  Arms: leptin repletion
Behavioral: Dietary modification — Subjects lose 10% of body weight via dietary restriction
  Other Names: no other name
Drug: T3 repletion — administer T3
  Other Names: no other name
  Arms: T3 repletion

SUMMARY:
Our previous studies have demonstrated that there is substantial metabolic opposition to the maintenance of an altered body weight. Leptin is a protein secreted by fat cells and the circulating concentrations of leptin are directly proportional to fat mass. Leptin-deficiency is associated with severe obesity in rodents and in humans and the obesity is relieved by leptin administration. These studies examine the hypothesis that some of this metabolic opposition cto the maintenance of an altered body weight can be relieved by restoring circulating concentrations of the hormone leptin to the same range as at usual body weight in subjects who are maintaining a reduced body weight. The basic design of this study is to observe subjects at a 10% reduced body weight and then again at that reduced body weight while receiving physiological leptin or T3 supplementation.

DETAILED DESCRIPTION:
We demonstrated a substantial metabolic resistance to maintenance of altered body weight. Leptin is secreted by fat cells in circulating concentrations that are directly proportional to fat mass. Leptin-deficiency is associated with severe obesity in rodents and in humans and the obesity is relieved by leptin administration. These studies examine the hypothesis that some of this metabolic opposition cto the maintenance of an altered body weight can be relieved by restoring circulating concentrations of the hormone leptin to the same range as at usual body weight in subjects who are maintaining a reduced body weight. The basic design of this study is to observe subjects at a 10% reduced body weight and then again at that reduced body weight while receiving physiological leptin or T3 supplementation.

ELIGIBILITY:
Healthy

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2000-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Effects of leptin repletion on hypometabolism/hyperphagia following weight loss | 9 months per subject
  Subjects are studied at usual weight and during maintenance of a 10% weight reduction while receiving either leptin repletion or a placebo in a single blind crossover design.

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia Presbyterian Medical Center, New York, New York, United States